CLINICAL TRIAL: NCT05131308
Title: Comparison of the Efficacy of Successful Leak Closure Between Available Leak Closure Methods for Clinically Relevant and Persisting Leaks Arising After Incomplete LAAC: Insights From the LAA-Leak Registry
Brief Title: Multimodality Evaluation of LAA Leaks Arising After Incomplete LAAC: Insights From the LAA-Leak Registry
Status: Completed | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-LAA Leak Registry-0007
Record Dates: First submitted 2021-10-26; First posted 2021-11-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Left Atrail Appendage Closure: Peri-device Leaks
Keywords: Left Atrial Appendage Closure; Central or peri-device leaks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Detachable embolization coils group: Patients who have an intervention for leak closure with detachable embolization coils
  Interventions: Other: leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA
- Vascular plugs/septal occluders group: Patients who have an intervention for leak closure with vascular plugs/CSO
  Interventions: Other: leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA
- RF Ablation group: Patients who have an intervention for leak closure with Radio Frequency Ablation (RFA)
  Interventions: Other: leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA

INTERVENTIONS:
Other: leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA — All patients were evaluated and followed with imaging, and per investigators' respective clinical judgement, then proceeded to have an intervention for leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA.

SUMMARY:
Closure of peri-device leaks (PDL) after incomplete LAAC have shown early feasibility, however no comparison study of all the leak closure modalities exists. Therefore, this is an attempt to report the first 3-way observational comparison study to date, with results in 160 total patients in 3 arms including detachable embolization coils, vascular plugs/septal occluders and Radiofrequency ablation.

DETAILED DESCRIPTION:
Left Atrial Appendage (LAA) Closure (LAAC) is a potent technique of LAA isolation and exclusion for stroke prevention in patients with atrial fibrillation, with evidence from the PROTECT-AF and PREVAIL-AF trials, including their 5-year follow-up assessments, solidifying LAAC as a viable option in these patients with comparable stroke reduction in comparison to oral anticoagulation (OAC) as well as a reduction in bleeding risk, hemorrhagic CVA, and mortality. However, the surge in the multiple methods of LAA exclusion has also brought to attention postprocedural complications specific to LAAC, namely, peri-device leaks (PDL). The stroke implication and classification of PDL itself still lacks consensus, with an increased thromboembolic (TE) potential due to PDL seen in patients with LARIAT and surgical ligation procedures, yet no statistically significant relationship seen in percutaneous and endocardial LAA closure approaches. PDL > 5mm has been widely accepted as clinically significant, although there remains limited data with no current established guidelines. Placement of a septal occluder device such as Amplatzer Vascular Plug, Detachable embolization coils, Gore Cardioform Septal Occluder (CSO; W.L. Gore and Associates, Newark DE), and radiofrequency ablation (RFA) have all emerged as options to resolve residual PDL and post-surgical/ligation leaks. However, there exists no head-to-head comparison between these modalities. Given their emergence, this is a proposed a multi-center observational study to further assess and evaluate these three treatment modalities for their efficacy for leak closure, assessment of pre-, peri- and post-procedural characteristics after leak closure, TE events, and bleeding risk, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at risk for stroke or thromboembolism that demonstrated any degree of the significant leak on follow up TEE imaging at least 4-6 weeks following either epicardial, endocardial, or surgical LAAC
2. Patients undergoing any form of eccentric or centric/central leak closure with available modalities (detachable embolization coils, vascular plus/septal/ASD occluders, or RF Ablation). Criteria for this was made based on the judgement of the operator, with no specific cutoffs for leak size, follow-up time from LAAC to leak closure, etc)
3. Age greater than 18 years

Exclusion Criteria:

1. Patients not undergoing leak closure after incomplete LAAC
2. Patients unable to complete 45 day follow-up imaging for reevaluation of LAA leak
3. Patients unable to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients at risk for stroke or thromboembolism that demonstrated any degree of the significant leak on follow up TEE imaging at least 4-6 weeks following either epicardial, endocardial, or surgical LAAC were included in this study population. All patients were evaluated and followed with imaging, and per investigators' respective clinical judgement, then proceeded to have an intervention for leak closure with either detachable embolization coils, vascular plugs/CSO, or RFA.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-01-11 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share the data

REFERENCES:
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Background] Nguyen A, Gallet R, Riant E, Deux JF, Boukantar M, Mouillet G, Dubois-Rande JL, Lellouche N, Teiger E, Lim P, Ternacle J. Peridevice Leak After Left Atrial Appendage Closure: Incidence, Risk Factors, and Clinical Impact. Can J Cardiol. 2019 Apr;35(4):405-412. doi: 10.1016/j.cjca.2018.12.022. Epub 2018 Dec 21. PMID 30935631
- [Background] Sahore A, Della Rocca DG, Anannab A, Mohanty S, Akella K, Murtaza G, Trivedi C, Gianni C, Chen Q, Bassiouny M, Ahmadian-Tehrani A, Macdonald B, Al-Ahmad A, Tarantino N, Cirone D, Horton RP, Romero J, Lakkireddy D, Di Biase L, Natale A. Clinical Implications and Management Strategies for Left Atrial Appendage Leaks. Card Electrophysiol Clin. 2020 Mar;12(1):89-96. doi: 10.1016/j.ccep.2019.11.010. PMID 32067651
- [Background] Albaghdadi, M., et al., Peri-Device Leaks after Percutaneous Left Atrial Appendage Closure: Clinical Significance and Unmet Diagnostic Needs. Structural Heart, 2020. 4(6): p. 475-481
- [Background] Mohanty S, Gianni C, Trivedi C, Gadiyaram V, Della Rocca DG, MacDonald B, Horton R, Al-Ahmad A, Gibson DN, Price M, Krumerman AK, Palma EC, Di Biase L, Lakkireddy D, Natale A. Risk of thromboembolic events after percutaneous left atrial appendage ligation in patients with atrial fibrillation: Long-term results of a multicenter study. Heart Rhythm. 2020 Feb;17(2):175-181. doi: 10.1016/j.hrthm.2019.08.003. Epub 2019 Aug 7. PMID 31400519
- [Background] Aryana A, Singh SK, Singh SM, O'Neill PG, Bowers MR, Allen SL, Lewandowski SL, Vierra EC, d'Avila A. Association between incomplete surgical ligation of left atrial appendage and stroke and systemic embolization. Heart Rhythm. 2015 Jul;12(7):1431-7. doi: 10.1016/j.hrthm.2015.03.028. Epub 2015 May 18. PMID 25998141
- [Background] Turagam MK, Velagapudi P, Kar S, Holmes D, Reddy VY, Refaat MM, Di Biase L, Al-Ahmed A, Chung MK, Lewalter T, Edgerton J, Cox J, Fisher J, Natale A, Lakkireddy DR. Cardiovascular Therapies Targeting Left Atrial Appendage. J Am Coll Cardiol. 2018 Jul 24;72(4):448-463. doi: 10.1016/j.jacc.2018.05.048. Epub 2018 Jun 26. PMID 29954658
- [Background] Jang SJ, Wong SC, Mosadegh B. Leaks after Left Atrial Appendage Closure: Ignored or Neglected? Cardiology. 2021;146(3):384-391. doi: 10.1159/000513901. Epub 2021 Mar 18. PMID 33735867
- [Background] Della Rocca DG, Horton RP, Di Biase L, Bassiouny M, Al-Ahmad A, Mohanty S, Gasperetti A, Natale VN, Trivedi C, Gianni C, Burkhardt JD, Gallinghouse GJ, Hranitzky P, Sanchez JE, Natale A. First Experience of Transcatheter Leak Occlusion With Detachable Coils Following Left Atrial Appendage Closure. JACC Cardiovasc Interv. 2020 Feb 10;13(3):306-319. doi: 10.1016/j.jcin.2019.10.022. Epub 2020 Jan 15. PMID 31954677
- [Background] Della Rocca DG, Horton RP, Tarantino N, Van Niekerk CJ, Trivedi C, Chen Q, Mohanty S, Anannab A, Murtaza G, Akella K, Gianni C, Bassiouny M, Ahmadian-Tehrani A, Al-Ahmad A, Burkhardt JD, Natale VN, Price M, Gallinghouse GJ, Gibson DN, Lakkireddy D, Di Biase L, Natale A. Use of a Novel Septal Occluder Device for Left Atrial Appendage Closure in Patients With Postsurgical and Postlariat Leaks or Anatomies Unsuitable for Conventional Percutaneous Occlusion. Circ Cardiovasc Interv. 2020 Oct;13(10):e009227. doi: 10.1161/CIRCINTERVENTIONS.120.009227. Epub 2020 Sep 18. PMID 32942913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between 2015 and 2021 in the US.
Period: Overall Study
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group
Started | 64 | 36 | 60
Completed | 64 | 36 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group | Total
Number analyzed (Participants) | 64 | 36 | 60 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (9.8) | 71.4 (7.2) | 76 (7.2) | 72.2 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 0 | 33 | 46
  Male | 51 | 36 | 27 | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Vascular Disease [Count of Participants; unit: Participants] | 33 | 18 | 15 | 66
History of CVA/TIA [Count of Participants; unit: Participants] | 21 | 12 | 24 | 57
TIA/CVA after primary LAAC before leak closure [Count of Participants; unit: Participants] | 9 | 3 | 6 | 18
Previous major bleeding [Count of Participants; unit: Participants]
  Intracranial hemorrhage | 7 | 4 | 6 | 17
  Gastrointestinal | 11 | 9 | 23 | 43
  No previous major bleeding | 46 | 23 | 31 | 100
Leak size prior to closure [Count of Participants; unit: Participants]
  Mild (1-2 mm) | 0 | 0 | 1 | 1
  Moderate (3-4 mm) | 23 | 27 | 16 | 66
  Severe (>5 mm) | 41 | 9 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Size of PDL After Leak Closure Procedure
Description: Size of leak in mm on TEE after leak closure procedure, immediately at the end of the procedure and at 1 year follow-up
Time Frame: Immediate postprocedural and 1 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group
Number analyzed (Participants) | 64 | 36 | 60
Participants
  Size of PDL immediately at the end of the procedure: Leak size - 0 mm | 0 | 0 | 0
  Size of PDL immediately at the end of the procedure: Leak size - < 1 mm | 64 | 36 | 60
  Size of PDL immediately at the end of the procedure: Leak size - 2-3 mm | 0 | 0 | 0
  Size of PDL immediately at the end of the procedure: Leak size - > 3 mm | 0 | 0 | 0
  Size of PDL at 1 year follow-up: Leak size - 0 mm | 45 | 36 | 31
  Size of PDL at 1 year follow-up: Leak size - < 1 mm | 10 | 0 | 19
  Size of PDL at 1 year follow-up: Leak size - 2-3 mm | 9 | 0 | 10
  Size of PDL at 1 year follow-up: Leak size - > 3 mm | 0 | 0 | 0

2. Secondary Outcome: Periprocedural Complications Occurring From Postoperative Day 0 - Day 7
Description: Periprocedural complications occurring from Postoperative days 0 - 7, including: device-related thrombus, pericardial effusion/pericardial tamponade requiring intervention and CVA.
Time Frame: From postoperative day 0 to day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group
Number analyzed (Participants) | 64 | 36 | 60
Participants
  Pericardial effusion/tamponade | 2 | 0 | 0
  Device-related thrombosis | 0 | 0 | 0
  CVA | 0 | 0 | 0
  Death | 0 | 0 | 0
  Vascular complications | 0 | 0 | 0
  No complications | 62 | 36 | 60

3. Secondary Outcome: Delayed Procedure-related Complications at 1 Year Follow-up
Description: Secondary Safety Endpoint: Delayed procedure-related complications at 1 year follow-up including device-related thrombus, pericardial effusion/ pericardial tamponade requiring intervention and CVA.
Time Frame: 1 year after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group
Number analyzed (Participants) | 64 | 36 | 60
Participants
  Pericardial effusion/tamponade | 0 | 0 | 0
  DRT | 0 | 0 | 0
  CVA | 0 | 0 | 0
  Death | 0 | 0 | 0
  Vascular complications | 0 | 0 | 0
  No complications | 64 | 36 | 60

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Detachable Embolization Coils Group | Vascular Plugs/Septal Occluders Group | RF Ablation Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/36 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/36 | 0/60
Other Adverse Events (participants affected / at risk) | 0/64 | 0/36 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT05131308/Prot_SAP_000.pdf